CLINICAL TRIAL: NCT00567294
Title: Improving Medication Adherence for Osteoporosis: A Community-Based Randomized Controlled Trial
Brief Title: Evaluating Ways to Improve Medication Use Among People With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Daniel H. Solomon, M.D.,MPH, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P60AR047782 (NIH); P60AR047782 (NIH); P60AR047782-06A1 (NIH)
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Medication adherence; Telephonic education; Motivational interviewing
MeSH Terms: conditions — Osteoporosis; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): Participants will receive mailed education materials on osteoporosis and medication use.
  Interventions: Behavioral: Mailed education
- B (Experimental): Participants will receive a telephone coaching program.
  Interventions: Behavioral: Telephone coaching program for patients
- C (Experimental): Participants will receive a telephone coaching program, and doctors of these participants will receive medication adherence alert notifications.
  Interventions: Behavioral: Telephone coaching program for patients; Behavioral: Medication adherence alert program for doctors

INTERVENTIONS:
Behavioral: Mailed education — Mailed education materials on osteoporosis and medication use over a 1-year period
  Arms: A
Behavioral: Telephone coaching program for patients — A telephone coaching program that will involve twelve monthly 5- to 10-minute phone calls from a health educator who is specially trained in osteoporosis. The phone calls will involve coaching participants on behavioral reinforcement strategies that will help them to continue taking their medications on schedule; phone calls will also include specially tailored education on osteoporosis and fracture prevention. A close family member or friend of the participant will also be contacted via phone two times during the study by the health educator. During these phone calls, the family member or friend will learn how to support the participant in such a way that medication adherence is more likely.
  Arms: B; C
Behavioral: Medication adherence alert program for doctors — Doctors of participants will receive written educational information on the rates of medication adherence, implications of nonadherence, and methods for improving adherence among people with osteoporosis. Doctors will also receive alerts on any patients who are not filling their medication prescriptions.
  Arms: C

SUMMARY:
Osteoporosis is a common bone disease in older adults in which the bones become weaker and prone to fracture. Medications are available to slow or even stop disease progression. However, very few adults who are prescribed osteoporosis medications actually follow through with filling their prescriptions and taking the medications. Ways to improve medication use have not been well developed or adequately tested. The purpose of this study is to evaluate a telephone coaching program, with or without helpful adherence notifications to doctors, in improving treatment adherence in older adults who are starting an osteoporosis medication.

DETAILED DESCRIPTION:
Fractures associated with osteoporosis are expected to rise to 3 million by 2025 with a cost of $25 billion in medical costs. Many of these fractures could be avoided through preventive measures, such as improved implementation of fall reduction strategies and use of effective medications. While medications can significantly reduce the chance of fractures among adults with osteoporosis, alarmingly few at-risk adults use osteoporosis treatments regularly. Only 10% to 30% of at-risk adults ever initiate osteoporosis medications, and of those, only 40% to 50% continue to fill their prescriptions after 1 year. There is a clear need to develop ways for improving adherence with osteoporosis medication regimens. The purpose of this study is to evaluate a telephone coaching program, with or without helpful adherence notifications to doctors, in improving treatment adherence in older adults who are starting an osteoporosis medication.

Participation in this study will last 1 year. Through random assignment of doctor practices, participants will fall into one of three groups.

* Group A participants will receive mailed education materials on osteoporosis and medication use throughout the 1-year study.
* Group B participants will receive monthly 5- to 10-minute phone calls from a health educator who is specially trained in osteoporosis. The phone calls will involve coaching participants on behavioral reinforcement strategies that will help them to continue taking their medications on schedule. Participants will also receive specially tailored education on osteoporosis and fracture prevention during the phone calls. A close family member or friend of the participant will be contacted via phone two times during the study year. During these phone calls, the family member or friend will learn how to support the participant in such a way that medication adherence is more likely.
* Group C participants will receive the same treatment as Group B. Doctors assigned to Group C will receive written educational information on the rates of medication adherence, implications of nonadherence, and methods for improving adherence among patients. Doctors will also receive alerts about any of their participating patients who are not filling medication prescriptions. The alert message will be provided in both paper and electronic format. The electronic format can be easily formatted, allowing the doctor to send a personalized letter to their patients.

At the end of the study, all participants will complete a mailed questionnaire on their behaviors and demographics. Doctors will complete a mailed questionnaire aimed at determining what parts of the interventions were well received. The occurrence of hip, forearm, and/or upper arm fractures will be evaluated using Medicare claims data.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the Pharmaceutical Assistance Contract for the Elderly (PACE) program at the Pennsylvania Department of Aging who begin taking a medication for osteoporosis

Exclusion Criteria:

* Unable to communicate over the telephone with health educators

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2087 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Medication adherence | At Month 12

SECONDARY OUTCOMES:
Medication persistence | At Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H. Solomon, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Timothy Gleeson, BS, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Solomon DH, Iversen MD, Avorn J, Gleeson T, Brookhart MA, Patrick AR, Rekedal L, Shrank WH, Lii J, Losina E, Katz JN. Osteoporosis telephonic intervention to improve medication regimen adherence: a large, pragmatic, randomized controlled trial. Arch Intern Med. 2012 Mar 26;172(6):477-83. doi: 10.1001/archinternmed.2011.1977. Epub 2012 Feb 27. PMID 22371876